CLINICAL TRIAL: NCT01547988
Title: Improving Balance Control and Self-Reported Lower Extremity Function in Community Dwelling Older Adults - A Randomized Control Study
Brief Title: Training Improves Balance Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRF 2001-056
Record Dates: First submitted 2012-02-29; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Accidental Falls
Keywords: Aging; Falls; Balance Control; Voluntary Step Execution Test; Dual-Task; Self-reported function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Training Intervention (Experimental): The Balance Training Intervention group received 24 training sessions over three months that included perturbation as well as dual-task exercises.
  Interventions: Other: Balance Training Intervention
- Reference Group (No Intervention)
  Interventions: Other: Balance Training Intervention

INTERVENTIONS:
Other: Balance Training Intervention — The intervention group participated in a total of 24 one-hour training sessions over a period of 12 weeks. The training program utilized different size balls as a general tool in a series of progressively more difficult exercises targeting sitting, standing, and gait-related balance control. The program included exercises at five different levels of progressively more challenging balance exercises. Levels 1-4 focused on voluntarily controlled balance exercises, whereas level 5 also included perturbation exercises to trigger automatic compensatory stepping responses. All levels included attention-demanding dual task exercises that required subjects to simultaneously perform motor and cognitive activities.

SUMMARY:
The purpose of this study was to evaluate the effect of a group-based functional and specific balance training program on balance function in healthy older adults. It is commonly considered difficult to improve balance function in healthy older adults. The program included dual-task exercises; physical training exercises and a cognitive task (e.g. reading or reciting a story) performed simultaneously, as well as perturbation exercises, where balance is challenged in unexpected ways.

The investigators hypothesized that following the proposed training, older adults would improve their speed of taking a step in both single and dual task conditions, refine their ability to control balance when standing still and improve their self-reported physical function.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Independently ambulatory (cane acceptable; not walker)
* Score better than 45 on the Berg Balance Scale
* Higher than 24 Mini-Mental Score

Exclusion Criteria:

* Severe focal muscle weakness or visual impairment
* Known neurological disorders (including stroke, Parkinson disease)
* Metastatic cancer
* Use of medication that impairs balance or strength

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2001-10; Primary Completion 2003-02 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Reaction time of dual task step execution | 12 weeks
  Subjects stand on a force platform and are asked to execute a step as rapidly as possible following a tactile stimulus on their heel while performing a cognitive attention demanding task (Stroop task - call out colors of words that are names of colors, e.g. the word "BLUE" is presented in yellow letters).

SECONDARY OUTCOMES:
Late Life Functional Disability Index - LLFDI | 12 weeks
  Self-reported measure of function

CONTACTS AND LOCATIONS:
Overall Officials: Lars IE Oddsson, PhD, Principal Investigator — NeuroMuscular Research Center, Boston University
Locations (1):
- NeuroMuscular Research Center, Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lars I. E. Oddsson, Patrick Boissy and Itshak Melzer. How to improve gait and balance function in elderly individuals-compliance with principles of training. European Review of Aging and Physical Activity Volume 4, Number 1, 15-23, DOI: 10.1007/s11556-007-0019-9
- [Background] Melzer I, Oddsson LI. The effect of a cognitive task on voluntary step execution in healthy elderly and young individuals. J Am Geriatr Soc. 2004 Aug;52(8):1255-62. doi: 10.1111/j.1532-5415.2004.52353.x. PMID 15271111
- [Background] Melzer I, Shtilman I, Rosenblatt N, Oddsson LI. Reliability of voluntary step execution behavior under single and dual task conditions. J Neuroeng Rehabil. 2007 May 29;4:16. doi: 10.1186/1743-0003-4-16. PMID 17535424